CLINICAL TRIAL: NCT05672693
Title: Study on the Accuracy of Intraocular Lens Calculation Formula
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-1059
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: the Accuracy of Intraocular Lens Calculation Formula

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Several Calculation Formulas of Intraocular Lens — Comparison of the accuracy of several intraocular lens calculation formulas

SUMMARY:
In this study, we will retrospectively collect patients who have performed phacoemulsification combined with intraocular lens implantation in our hospital, collect various preoperative biometric data and postoperative refractive data of patients, conduct statistical analysis, and compare the accuracy of various IOL calculation formulas.

ELIGIBILITY:
Inclusion Criteria:

* (1) Conform to the diagnosis of cataract; (2) No complications occurred during and after operation; (3) Before and after operation, the measurement of ocular biological characteristics and refractive state can be successfully completed; (4) Patients who can be followed up regularly after operation.

Exclusion Criteria:

* (1) Serious intraoperative or postoperative complications; (2) Complicated with other eye diseases unsuitable for intraocular lens implantation; (3) Patients with systemic diseases cannot tolerate surgery; (4) Patients with incomplete follow-up data.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were previously diagnosed as "senile cataract" in the Ophthalmology Center of the Second Affiliated Hospital of Zhejiang University Medical College and who performed "phacoemulsification cataract extraction combined with intraocular lens implantation"
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mean absolute error | 1 week、1 month and 3 months postoperation
  The Friedman test was applied to compare the median absolute error between the formulas after the zeroing of the mean numerical error.
  Post hoc analysis and Bonferroni correction was performed for multiple comparisons.

SECONDARY OUTCOMES:
Distribution of error within ± 0.25D, ± 0.5D, ± 0.75D,and ± 1.0D | 1 week、1 month and 3 months postoperation
  Frequency comparisons were made with the chi-square test

CONTACTS AND LOCATIONS:
Overall Officials: Wen Xu, Study Chair — Second Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No